CLINICAL TRIAL: NCT04563494
Title: The Effects of IV vs Oral Dexamethasone on Postoperative Nausea, Vomiting, Pain, and Drug Cost in Children Undergoing Tonsillectomy: A Randomized Controlled Prospective Non-inferiority Study
Brief Title: The Effects of IV vs Oral Dexamethasone on Postoperative Nausea, Vomiting, and Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-1742
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IV Dexmethsone and oral placebo (Active Comparator)
  Interventions: Drug: dexamethasone
- Oral dexamethasone and IV placebo (Active Comparator)
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — Prevention of post op nausea and vomiting

SUMMARY:
The hypothesis being tested in this study is that perioperative oral administration of dexamethasone, when compared to intravenous (IV) administration, offers a similar reduction in postoperative nausea and vomiting (PONV), and reduction in postoperative pain in pediatric patients undergoing tonsillectomy with or without adenoidectomy and/or tympanostomy tube placement. The specific aim of this study is to demonstrate non-inferiority of oral dexamethasone when compared to IV dexamethasone, given that there is currently a severe, sudden, and world-wide shortage of IV dexamethasone given its recent use in treating patients with covid19 disease.

DETAILED DESCRIPTION:
written consent, patients will be randomized at the time of arrival to the preoperative care center on the day of surgery. One hundred twenty-six patients, 3 to 7 years of age undergoing tonsillectomy with or without adenoidectomy and tympanostomy tube placement, will be included in this study. Children who received antiemetics, steroids, anti-histaminic, or psychoactive drugs during the week before surgery will be excluded. Patients will be prospectively randomized to receive oral or IV dexamethasone 0.5 mg/kg (maximum dose 8 mg). Patients in the IV group will receive the dose once an IV is placed in the operating room. They will receive an oral placebo once consent is obtained on arrival to the preoperative center on the day of surgery. Patients in the oral group will receive their dose once consent is obtained on arrival to the preoperative center on the day of surgery. They will receive a placebo once the IV is placed in the operating room. Randomization will be via a computer-generated table of numbers. Study drugs will be marked only with a coded number label. The anesthesiologist, surgeon, patient, and family will be unaware of drug identity. All medication preparation and handling will be done by CHCO Investigational Drug Service.

Patients will be fasted for solid foods for eight hours before surgery; clear liquids will be permitted until two hours before surgery. A standard anesthetic technique will be used. Premedication with oral acetaminophen 12.5-15 mg/kg will be given on arrival to the preoperative center. After obtaining consent study drug or placebo will be given at least 20 minutes before surgery. General anesthesia will be induced with sevoflurane and 60% nitrous oxide in oxygen via mask followed by insertion of an intravenous (IV) cannula. Dexamethasone or placebo will be given immediately following IV placement. Propofol 2 mg/kg and fentanyl 1 µg/kg will be given to facilitate intubation. Anesthesia will be maintained with a mixture of sevoflurane and air (FiO2 < 0.3All children will receive fentanyl 1-3 µg/kg (titrated to pain response in the operating room) and dexmedetomidine 0.5 µg/kg once surgery starts. All children will receive ondansetron 0.1 mg/kg (maximum dose 4 mg).All children will receive 20 mL/kg lactated Ringer's solution during surgery (maximum IV fluid 750 mL given short time of surgical procedure). Routine monitoring including heart rate (ECG), arterial oxygen saturation (SpO2), blood pressure, temperature and end-tidal CO2 will be used throughout surgery. Surgical technique will be standardized, and all patients will have their stomachs suctioned at the completion of surgery.

Each subject will be assessed by nursing staff utilizing standard of care practices in the PACU and patients will stay in the PACU (phase one and two) for 4 hours after surgery. Postoperative nausea and vomiting (PONV) will be defined as vomiting and/or retching without expulsion of gastric content and will be treated with IV phenergan (0.25 mg/kg, maximum 25 mg) followed, if necessary, by IV diphenhydramine (1 mg/kg maximum 50 mg). Pain will be assessed using the numeric pain scale 0-10, Faces, Legs, Arms, Crying, Consolability Scale (FLACC Scale), or Revised Faces Scale.12,13 Pain scores > 5 will be treated with IV fentanyl 0.5 µg/kg that can be repeated every 5 minutes for pain when necessary.

ELIGIBILITY:
Inclusion Criteria:

* 3-7 years of age
* tonsillectomy with or without adenoidectomy and tympanostomy tube placement

Exclusion Criteria:

* Subjects receiving one week before surgery:

  •-antiemetics
* steroids
* anti-histaminic
* psychoactive drugs

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of post op nausea and vomiting | 4 hours
  post-op nausea and vomiting as evidenced by vomiting and/or retching without expulsion of gastric content

SECONDARY OUTCOMES:
pain scores and surgical re-exploration for bleeding | 4 hours
  Pain as evidenced by a numeric pain scale 0-10, Faces, Legs, Arms, Crying, Consolability Scale (FLACC Scale), or Revised Faces Scale.12,13 .
  surgical re-exploration as evidenced by the return to O.R. for bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Brooks Peterson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No